CLINICAL TRIAL: NCT06583200
Title: End Expiratory Occlusion Test for Evaluation of Fluid Responsiveness in Comparison to Passive Leg Raising Test in Mechanically Ventilated Post Cardiac Surgery Patients
Brief Title: Fluid Responsiveness in Post Cardiac Surgery Patients
Acronym: Cardiac
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Screening
Other Study IDs: FAMSU MD 220/2022
Record Dates: First submitted 2024-08-03; First posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-04

CONDITIONS: Cardiac Complication
Keywords: Cardiac surgery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- End Expiratory Occlusion Test (Other): Pulse pressure variation before and after end expiratory occlusion test
  Interventions: Diagnostic Test: End Expiratory Occlusion Test; Diagnostic Test: Passive Leg Raising Test
- Passive leg raising test (Other): Pulse pressure variation before and after passive leg raising test
  Interventions: Diagnostic Test: End Expiratory Occlusion Test; Diagnostic Test: Passive Leg Raising Test

INTERVENTIONS:
Diagnostic Test: End Expiratory Occlusion Test — All studied mechanically ventilated patients under post operative sedation. EEO test will be applied to predict probable responder and probable non-responder according to pulse pressure variation in accordance to previous study where the response to volume expansion was defined as an increase in pulse pressure of 5% or more
Diagnostic Test: Passive Leg Raising Test — All studied mechanically ventilated patients under post operative sedation.Passive leg raising test will be applied to predict probable responder and probable non-responder according to the PPV in accordance to previous study where the response to volume expansion was defined as an increase in pulse pressure of at least 10%

SUMMARY:
The aim of the study is to compare end expiratory occlusion test to passive leg raising test for prediction of fluid responsiveness in post cardiac surgery mechanically ventilated patients.

DETAILED DESCRIPTION:
Circulatory hypervolemia and hypovolemia are both associated with worse outcomes.Intravenous fluids are similar to drugs, with serious adverse effects and changeful efficacy. Fluids should be administered only if indicated. Passive leg raising test transiently increase venous return which can be used to evaluate fluid responsiveness.There is growing evidence that the End expiratory occlusion (EEO) test reliably detects fluid responsiveness. In patients under mechanical ventilation, the inspiration increases intra-thoracic pressure and decreases venous return. The expiratory hold augments the cardiac preload which, in case of preload responsiveness, leads to a significant increase of cardiac output (CO).EEO prevents any variation in intra-thoracic pressure leading to an increase in venous return, cardiac preload and stroke volume in preload-responsive patients. There're no studies comparing EEO with passive leg raising test in cardiac surgery patients. So, this is the target of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age group: 21-60years old
* Sex: eligible both sexes
* Post cardiac surgery
* Sedated intubated mechanically ventilated patients (Controlled ventilation with no respiratory effort)

Exclusion Criteria:

* Patients refusal
* Pregnancy or any medical condition that may affect the intra abdominal pressure.
* Lower limb deep venous thrombosis Open chest conditions impaired left-ventricular ejection fraction (<45%), arrhythmias, inter-ventricular shunt, severe peripheral arterial occlusive disease and the need for intra-aortic balloon counter pulsation

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-12 (Estimated)

PRIMARY OUTCOMES:
Predictive value of EEO and passive leg raising | One year
  Predictive value of EEO and passive leg raising to fluid responsiveness in post cardiac surgery mechanically ventilated patients Pulse pressure variation before and after passive leg raising test

SECONDARY OUTCOMES:
Arterial blood pressure | One year
  Effect of EEO and passive leg raising to fluid responsiveness on arterial blood pressure in post cardiac surgery mechanically ventilated patients
Heart rate | One year
  Effect of EEO and passive leg raising to fluid responsiveness on heart rate in post cardiac surgery mechanically ventilated patients

OTHER OUTCOMES:
Central venous pressure | One year
  Effect of EEO and passive leg raising to fluid responsiveness on central venous pressure in post cardiac surgery mechanically ventilated patients

CONTACTS AND LOCATIONS:
Overall Officials: Marwa Khairy, Professor, Study Director — Ain Shams University
Locations (1):
- Faculty of medicine Ain Shams University, Cairo, Cairo Governorate, Egypt